CLINICAL TRIAL: NCT03366415
Title: Non-inferiority Prospective Randomized Trial Comparing Sequential Chemoradiotherapy With Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Sequential or Concurrent Chemoradiotherapy in Patients With Locoregionally Advanced NPC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaosu Hu (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Affiliated Hospital of Jiangnan University (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Chaosu Hu, chief physician, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP2017-02（SANDWICH）
Record Dates: First submitted 2017-12-02; First posted 2017-12-08 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; concurrent chemoradiotherapy; sequential chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin; Neoadjuvant Therapy; Chemotherapy, Adjuvant; Induction Chemotherapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Stratified by stage
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Induction chemotherapy+IMRT+adjuvant chemotherapy (Experimental): Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (25 mg/m² d1-3) every 3 weeks for 2 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), followed by gemcitabine (1000 mg/m² d1,8) and cisplatin (25 mg/m² d1-3) every 3 weeks for 2 cycles.
  Interventions: Drug: gemcitabine and cisplatin (Induction and adjuvant chemotherapy); Radiation: IMRT
- Induction chemotherapy+IMRT and concurrent cisplatin (Active Comparator): Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (25 mg/m² d1-3) every 3 weeks for 2 cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT), concurrently with cisplatin 30 mg/m² every week.
  Interventions: Drug: gemcitabine and cisplatin (Induction chemotherapy); Radiation: IMRT and concurrent cisplatin

INTERVENTIONS:
Drug: gemcitabine and cisplatin (Induction and adjuvant chemotherapy) — Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (25mg/m² d1-3) every 3 weeks for 2 cycles before IMRT and after IMRT.
  Arms: Induction chemotherapy+IMRT+adjuvant chemotherapy
Radiation: IMRT — Intensity modulated-radiotherapy (IMRT) is given as 2.2 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 or 70.4 Gy to the primary tumor
  Arms: Induction chemotherapy+IMRT+adjuvant chemotherapy
Drug: gemcitabine and cisplatin (Induction chemotherapy) — Patients receive gemcitabine (1000 mg/m² d1,8) and cisplatin (25mg/m² d1-3) every 3 weeks for 2 cycles before concurrent chemoradiotherapy.
  Arms: Induction chemotherapy+IMRT and concurrent cisplatin
Radiation: IMRT and concurrent cisplatin — Intensity modulated-radiotherapy (IMRT) is given as 2.2 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 or 70.4Gy to the primary tumor, concurrently with cisplatin 30mg/m² every week.
  Arms: Induction chemotherapy+IMRT and concurrent cisplatin

SUMMARY:
The purpose of this study is to compare the efficacy and safety of sequential chemoradiotherapy (induction chemotherapy + intensity-modulated radiotherapy +adjuvant chemotherapy) with induction chemotherapy plus concurrent chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma (NPC), in order to confirm the value of sequential chemoradiotherapy in NPC patients.

DETAILED DESCRIPTION:
Patients with non-keratinizing NPC III-IVA (UICC/AJCC 8th edition) are randomly assigned to receive sequential chemoradiotherapy (induction chemotherapy + intensity-modulated radiotherapy + adjuvant chemotherapy) or induction chemotherapy plus concurrent chemoradiotherapy. Intensity-modulated radiotherapy (IMRT) is given as 2.2 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 or 70.4 Gy to the primary tumor. The induction or adjuvant chemotherapy is given gemcitabine (1000 mg/m² d1,8) and cisplatin (25mg/m² d1-3) every 3 weeks for two cycles. The concurrent chemotherapy is given cisplatin 30 mg/m² every week concurrently with IMRT. Our primary endpoint is failure-free survival(FFS) and grade III mucositis during radiation. Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), distant failure-free survival (D-FFS) rates and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type)
* Tumor staged as III-IVA (according to the 8th AJCC edition).
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Age between 18 and 65 years old.
* Adequate marrow: Neutrophil count ≥2000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) ≤ 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ 1.5ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Evidence of distant metastasis
* Prior chemotherapy, radiotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Other previous or concomitant cancer.
* Pregnancy or lactation.
* Presence of an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, immune deficiency, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or emotional disturbance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3-year
  Failure-free survival is calculated from the date of randomisation to the date of treatment failure or death from any cause, whichever is first.
Grade III or more mucositis | From the start of radiotherapy to 30 days after radiotherapy
  Grade III or more mucositis during radiotherapy

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 3-year
  Locoregional failure-free survival is calculated from randomization to the first locoregional failure.
Distant failure-free survival | 3-year
  Distant failure-free survival is calculated from randomization to the first remote failure.
Short-term treatment response | Two weeks after completion of induction chemotherapy. Three months after completion of the radiotherapy.
  Treatment response after induction chemotherapy, IMRT and completion of treatment.
Number of participants with adverse events | up to 3 years
  Incidence of acute and late toxicity
Quality of Life | up to 3 years
  Use EORTC QLQ-HN35.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xue F, Ou D, Xie C, Lin S, Li J, Chen X, Zhang F, Ying H, Lu X, Shen C, Xu T, Ou X, Li W, Zhou X, Du C, Zhou C, Hu C, He X. Sequential vs Induction Plus Concurrent Chemoradiotherapy in Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA Oncol. 2025 Jul 24;11(9):1011-20. doi: 10.1001/jamaoncol.2025.2191. Online ahead of print. PMID 40705321